CLINICAL TRIAL: NCT06344897
Title: Effectiveness of Kinesio Tape Applied After Open Appendectomy Surgery in Children: Randomized Controlled Study
Brief Title: The Effect of Kinesio Taping in Pediatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Nigde Omer Halisdemir University (Other); University of Health Sciences Konya Health Application and Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: mac1
Record Dates: First submitted 2024-01-24; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-12

CONDITIONS: Appendicitis; Surgery; Pain, Acute
MeSH Terms: conditions — Appendicitis; Acute Pain

STUDY DESIGN:
Intervention Model Description: The effect of kinesio taping on pain in children aged 6-12 years who had open appendicitis surgery.
Who Masked: Participant
Masking Description: The research is in a parallel group, single-blind randomized controlled experimental design.
  Simple randomization will be applied to children who have had open appendicitis surgery and meet the inclusion criteria, without any stratification in the study.
  In order to determine which group the 68 children who meet the sample selection criteria in the study group will be included in, numbers from 1 to 68 will be randomly distributed to 2 groups through a computer program (https://www.randomizer.org/) without number repetition. 34 patients will be assigned to the experimental group and 34 patients to the control group. Since the person who will actively apply the taping in the study is the researcher, only the children will be blinded, therefore a single blind design will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Experimental): The taping process will be done immediately after appendicitis surgery. Kinesio taping will continue until child's first gas is released.
  In addition to the standard pain management applied in the clinic, Kinesio tape will be applied to children who have had appendicitis surgery.
  Interventions: Other: Kinesio taping
- Control group (No Intervention): The control group will receive standard pain treatment without any intervention. The group will not receive any other intervention.

INTERVENTIONS:
Other: Kinesio taping — After appendicitis surgery, children will receive Kinesio taping in addition to the standard pain management applied in the clinic.
  Arms: Kinesio Taping

SUMMARY:
This study was planned to determine the effect of kinesio taping (KT) applied to the abdominal area after surgery on pain and gas output in children aged 6-12 years who had open appendicitis surgery.

DETAILED DESCRIPTION:
It is stated that kinesio taping, alone or in combination, is an alternative application for the pain management of various disease and symptom processes. These sources state that kinesion relieves pain and makes movement easier. When the literature was examined, no study could be found examining the effectiveness of kinesio tape application in pain management and flatulence in the post-operative period in children who had appendicitis surgery. For this reason, this study aimed to examine the effect of kinesio taping applied to the abdominal area on pain and gas output after appendicitis surgery in children between the ages of 6-12.

ELIGIBILITY:
Inclusion Criteria:

* Open appendicitis surgery was performed,
* Are between the ages of 6-12,
* Conscious, literate and without hearing or speech problems,
* Children who do not have a mental disorder and agree to participate in the research will be included.

Exclusion Criteria:

* Exclusion Criteria:
* Do not apply analgesic treatment other than routine application.
* Patients who develop complications during the operation will be excluded from the study.
* Those with acute appendicitis or Angenesis appendicitis

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Kinesio tape applying affects pain in children aged 6-12 years who have appendicitis surgery. | up to 6-24 hours
  Visual Analog Scale (VAS): The scale is used to measure pain intensity. The scale consists of a horizontal or vertical ruler, 10 cm or 100 mm long, showing "no pain" at one end and "the most severe pain" possible at the other end. At the left end of the line is the expression "No pain" or "Pain is completely gone", while at the right end is the expression "Unbearable pain" or "There is no decrease in pain".
Kinesio tape applying affects fear in children aged 6-12 years who have appendicitis surgery. | up to 6-24 hours
  It is used to evaluate pain and anxiety in children before and during the procedure.The scale can also be scored by the parent and the researcher. The scale consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety).

SECONDARY OUTCOMES:
Kinesio taping affects gas output time in children aged 6-12 years who have appendicitis surgery | up to 6-24 hours
  When the Kinesio Taping ends, children's with appendicitis surgery the Gas exit time will decrease.
  1-Gas Exit Form This form consists of two parts. The first part is where the child's surgery discharge time is written. The second part is where the time of the first gas exist is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim AKKOYUN, Assoc.Prof., Study Chair — University of Health Sciences Konya Health Application and Research Center; Bayram Sonmez UNUVAR, Ph.D., Principal Investigator — KTO Karatay University; Hilal KURT SEZER, Ph.D., Principal Investigator — Niğde Ömer Halisdemir University; Muzaffer ERDOĞAN, Md., Principal Investigator — University of Health Sciences Konya Health Application and Research Center; Sabit DERE, Md., Principal Investigator — University of Health Sciences Konya Health Application and Research Center; Merve ASKIN CERAN, M.Sc., Principal Investigator — KTO KaratayUniversity
Locations (1):
- University of Health Sciences Konya Health Application and Research Center, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Atalan Efkere P, Tarsuslu T. The effects of Kinesio taping on static and dynamic balance in children with down syndrome: a randomized controlled trial. Somatosens Mot Res. 2024 Jun;41(2):115-122. doi: 10.1080/08990220.2023.2183829. Epub 2023 Feb 28. PMID 36852775
- [Background] Gerçeker, G., Ayar, D., Özdemir, Z., & Bektaş, M. (2018). Çocuk anksiyete skalası-durumluluk ve çocuk Korku ölçeğinin Türk diline kazandırılması. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 11(1), 9-13.
- [Background] Mohamed RA, Yousef AM, Radwan NL, Ibrahim MM. Efficacy of different approaches on quality of upper extremity function, dexterity and grip strength in hemiplegic children: a randomized controlled study. Eur Rev Med Pharmacol Sci. 2021 Sep;25(17):5412-5423. doi: 10.26355/eurrev_202109_26648. PMID 34533816
- [Background] Ortiz Ramirez J, Perez de la Cruz S. Therapeutic effects of kinesio taping in children with cerebral palsy: a systematic review. Arch Argent Pediatr. 2017 Dec 1;115(6):e356-e361. doi: 10.5546/aap.2017.eng.e356. English, Spanish. PMID 29087112
- [Background] Parmar ST, Dhanuka HR, Shetty DR. Effectiveness of Kinesio Taping and Exercises for Pronated Feet in Children with Neurodevelopmental Disorders: A Cross Over Study. Niger J Clin Pract. 2022 Jan;25(1):21-26. doi: 10.4103/njcp.njcp_62_21. PMID 35046190